CLINICAL TRIAL: NCT01437813
Title: Bioavailability of Glimepiride/Extended Release Metformin (4/850 mg) After a High Fat Diet, in Healthy Mexican Volunteers
Brief Title: BIOAVAILABILITY OF Glimepiride/Extended Release Metformin (GLI/METXR): High Fat Diet Study
Acronym: GLMT13
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Collaborators: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLMT13-SIL
Record Dates: First submitted 2011-09-19; First posted 2011-09-21 (Estimated); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Healthy
Keywords: DM2; glimepiride; metformin extended release
MeSH Terms: interventions — glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Group A: Glimepiride / Extended Release Metformin (Experimental): Pharmaceutical Form: Tablets Dosage: 4 mg / 850 mg Administration way: Oral
  Interventions: Drug: Glimepiride/ Extended release Metformin

INTERVENTIONS:
Drug: Glimepiride/ Extended release Metformin — One tablet of Glimepiride/metformin extended release (4/850 mg) was administered as a single oral dose. Patients received a high fat diet 30 min before administration.
  Other Names: GLIMETXR

SUMMARY:
Objective:

The purpose of this study is to evaluate the effect of food intake in bioavailability (BA) of the combination Glimepiride/ extended release Metformin GLI/METXR (4/850mg) in healthy Mexican volunteers.

Methods: A prospective, longitudinal, open label, non randomized study, was performed. A single oral dose of GLI/METXR (4/850 mg) was administered to 24 health Mexican volunteers 30 min after a high fat meal.

DETAILED DESCRIPTION:
Blood samples were collected before the administration and 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6.7, 8, 10, 12, 16, 20, 24 and 30 hours post-administration. Plasma concentration of the drug was measured by using HPLC. Plasma concentration of both drugs were measured using high-performance liquid chromatography (HPLC). Plasma concentration time curves were plotted for each volunteers, and pharmacokinetic parameters (PK) were calculated. The pharmacokinetic parameters to be determined are: Cmax, Tmax, AUC0-t, AUC0-inf, TMR, Ke, T1 / 2 of glimepiride and metformin. The statistical analysis will be descriptive for plasma concentrations with respect to time and the pharmacokinetic parameters of Cmax, Tmax, AUC0-t, AUC0-inf, TMR, Ke, T1/2 of glimepiride and metformin. Adverse events were determined using clinical and laboratory test results throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Mexican volunteers, considered healthy according to standard screening assessments
* Aged between 18 and 50 years old
* Body mass index (BMI) was 18 to 27.5

Exclusion Criteria:

* Those with a history or evidence of cardiovascular, renal, hepatic, gastrointestinal, neurologic, muscular, metabolic, or hematologic abnormality
* Any acute or chronic disease
* Any drug allergy and female volunteers positive to urinary pregnancy test or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-01; Primary Completion 2011-01 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Profile | Predose,0.25, 0.5, 0.75, 1, 1.5, 2, 2.5,3, 3.5, 4, 4.5, 5, 6, 7, 8, 10, 12, 16,20, 24 y 30 hours post-dose
  Cmax, Area Under Curve, Tmax

SECONDARY OUTCOMES:
Adverse Events | 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5,3, 3.5, 4, 4.5, 5, 6, 7, 8, 10, 12, 16,20, 24 y 30 hours post-dose
  Any change in health or undesirable experience in volunteers related or unrelated with the experimental drug.
  Adverse events were determined using clinical and laboratory test results, throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Yamanqui Ibañez, Dr., Principal Investigator — INVESTIGACIÓN FARMACOLÓGICA Y BIOFARMACEUTICA.
Locations (1):
- Investigación Farmacológica Y Biofarmaceutica, S.A. de C.V., México, Mexico

REFERENCES:
- [Result] Badian M, Korn A, Lehr KH, Malerczyk V, Waldhausl W. Determination of the absolute bioavailability of glimepiride (HOE 490), a new sulphonylurea. Int J Clin Pharmacol Ther Toxicol. 1992 Nov;30(11):481-2. No abstract available. PMID 1490793
- [Result] Bailey CJ, Turner RC. Metformin. N Engl J Med. 1996 Feb 29;334(9):574-9. doi: 10.1056/NEJM199602293340906. No abstract available. PMID 8569826
- [Result] Campbell RK. Glimepiride: role of a new sulfonylurea in the treatment of type 2 diabetes mellitus. Ann Pharmacother. 1998 Oct;32(10):1044-52. doi: 10.1345/aph.17360. PMID 9793597
- [Result] Davidson MB, Peters AL. An overview of metformin in the treatment of type 2 diabetes mellitus. Am J Med. 1997 Jan;102(1):99-110. doi: 10.1016/s0002-9343(96)00353-1. PMID 9209206
- [Result] DeFronzo RA. Pharmacologic therapy for type 2 diabetes mellitus. Ann Intern Med. 1999 Aug 17;131(4):281-303. doi: 10.7326/0003-4819-131-4-199908170-00008. PMID 10454950